CLINICAL TRIAL: NCT04325763
Title: A Randomized, Double-blind and Imitation, Placebo Parallel Control, Multicentre Phase III Study of TQB2450 With or Without Anlotinib as Consolidation Treatment in Subjects With Locally Advanced/Unresectable (Stage III) Non-Small Cell Lung Cancer That Have Not Progressed After Prior Concurrent/Sequential Chemoradiotherapy
Brief Title: A Study of TQB2450 in Subjects With Stage III Non-Small Cell Lung Cancer(NSCLC)
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TQB2450-III-05
Record Dates: First submitted 2020-03-25; First posted 2020-03-30 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Stage III Non-small-cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — anlotinib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- TQB2450+Anlotinib (Experimental): TQB2450 1200 mg administered intravenously (IV) on Day 1 of each 21-day cycle ,Anlotinib capsules 8 mg given orally, once daily in 21-day cycle (14 days on treatment from Day 1-14, 7 days off treatment from Day 15-21).
  Interventions: Drug: TQB2450; Drug: Anlotinib
- TQB2450+Anlotinib(blank) (Experimental): TQB2450 1200 mg administered intravenously (IV) on Day 1 of each 21-day cycle ,Anlotinib capsules 0 mg given orally, once daily in 21-day cycle (14 days on treatment from Day 1-14, 7 days off treatment from Day 15-21).
  Interventions: Drug: TQB2450; Drug: Anlotinib(blank)
- TQB2450(blank)+Anlotinib(blank) (Placebo Comparator): TQB2450 0 mg administered intravenously (IV) on Day 1 of each 21-day cycle ,Anlotinib capsules 0 mg given orally, once daily in 21-day cycle (14 days on treatment from Day 1-14, 7 days off treatment from Day 15-21).
  Interventions: Drug: TQB2450(blank); Drug: Anlotinib(blank)

INTERVENTIONS:
Drug: TQB2450 — TQB2450 is a humanized monoclonal antibody targeting programmed death ligand-1 (PD-L1), which prevents PD-L1 from binding to PD-1 and B7.1 receptors on T cell surface, restores T cell activity, thus enhancing immune response and has potential to treat various types of tumors.
  Arms: TQB2450+Anlotinib; TQB2450+Anlotinib(blank)
Drug: Anlotinib — a multi-target receptor tyrosine kinase inhibitor
  Arms: TQB2450+Anlotinib
Drug: TQB2450(blank) — Subjects administrated TQB2450 (blank) intravenously (IV) on Day 1 of each 21-day
  Arms: TQB2450(blank)+Anlotinib(blank)
Drug: Anlotinib(blank) — Subjects administrated anlotinib (blank) in fasting conditions, once daily in 21-day cycle (14 days on treatment from Day 1-14, 7 days off treatment from Day 15-21)
  Arms: TQB2450(blank)+Anlotinib(blank); TQB2450+Anlotinib(blank)

SUMMARY:
This study is a randomized, double-blind, double-dummy,placebo parallel controlled, multi-centre,phase III clinical trial to evaluate the efficacy and safety of TQB2450 with or without anlotinib compared with placebo as consolidation treatment in subjects with locally advanced/unresectable (Stage III) Non-Small Cell Lung Cancer that has not progressed after prior concurrent/sequential chemoradiotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. 18-75 years old ; Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1; Life expectancy ≥ 3 months.
2. Histologically or cytologically confirmed unresectable (Stage III) Non-Small Cell Lung Cancer.
3. At least has one measurable lesion before radiotherapy.
4. At least has one type of platinum-containing chemotherapy, Absence of progression after concurrent/sequential chemoradiotherapy.
5. Adequate laboratory indicators.
6. No pregnant or breastfeeding women, and a negative pregnancy test.
7. Understood and signed an informed consent form.

Exclusion Criteria:

1. Squamous cell carcinoma meets following conditions should be excluded:

   1. Cavernous lung cancer.
   2. Has hemoptysis and maximum daily hemoptysis volume ≥ 2.5ml within 1 month before the first administration.
2. Has received anti-angiogenic drugs or other PD-1 / PD-L1 / CTLA-4 antibody therapy or other immunotherapy against PD-1 / PD-L1 / CTLA-4.
3. Severe hypersensitivity occurs after administration of other monoclonal antibodies.
4. Diagnosed and/or treated additional malignancy within 5 years with the exception of cured basal cell carcinoma of skin ,carcinoma in situ of prostate,and carcinoma in situ of cervix.
5. Pathologically confirmed mixed small cell and non-small cell lung cancer.
6. EGFR gene mutations.
7. Has any active autoimmune disease or history of autoimmune disease.
8. After the early stage of chemoradiotherapy, the treatment toxicity ≥ grade 2 is not fully alleviated.
9. Has ≥grade 2 pneumonia.
10. Immunosuppressant or systemic or absorbable local hormone therapy is required to achieve the aim of immunosuppression (dose > 10mg/ day prednisone or other therapeutic hormones) and is still used within 2 weeks after the first administration.
11. Has multiple factors affecting oral medication.
12. Has active bleeding or a persistent decrease in hemoglobin.
13. Has any bleeding or bleeding events ≥grade 3 in the first 4 weeks before the first administration.

2.Has received anti-angiogenic drugs or other PD-1 / PD-L1 / CTLA-4 antibody therapy or other immunotherapy against PD-1 / PD-L1 / CTLA-4.

14. Has unhealed wounds, fractures, active gastric and duodenal ulcers, positive continuous fecal occult blood, ulcerative colitis in the first 4 weeks before the first administration.

15. Has received NMPA approved anti-tumor drugs or immunomodulatory drugs for systemic treatment within 2 weeks before the first administration.

16.Has a history of a hematological system transplantation or organ transplantation.

17. Has active diverticulitis、peritoneal abscess, intestinal obstruction. 18. Has any serious and/or uncontrollable disease. 19. According to the judgement of the investigators, there are other factors that may lead to the termination of the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 315 (Estimated)
Dates: Start 2020-05-27 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) evaluated by Independent Review Committee(IRC) | up to 33 months
  PFS defined as the time from randomization until the first documented progressive disease (PD) or death from any cause, based on IRC.

SECONDARY OUTCOMES:
PFS evaluated by Investigator | up to 33 months
  PFS defined as the time from randomization until the first documented progressive disease (PD) or death from any cause, based on investigator.
Overall survival (OS) | up to 5 years
  OS defined as the time from randomization to death from any cause. Participants who do not die at the end of the extended follow-up period, or were lost to follow-up during the study, were censored at the last date they were known to be alive.
Overall response rate (ORR) | up to 33 months
  Percentage of participants achieving complete response (CR) and partial response (PR).
Disease control rate（DCR） | up to 33 months
  Percentage of participants achieving complete response (CR) and partial response (PR) and stable disease (SD).
Duration of response（DOR） | up to 33 months
  The time when the participants first achieved complete or partial remission to disease progression.
PFS rate at month 6 | up to 6 months
  The percentage of PFS at month 6
PFS rate at month 12 | up to 12 months
  The percentage of PFS at month 12
Biomarkers, such as PD-L1 expression, etc. | up to 33 months
  Tissue samples were collected during the screening period for pd-l1 analysis. Blood samples were collected for Tumor Mutation Burden (TMB) test before enrollment (within 7 days before medication) and after exit (±3 days).
Immunogenicity, such as the incidence of ADA | on day 1, 42, 105, 189 and 90 days after the last administration.
  Degree of the immune response caused by the drug.

CONTACTS AND LOCATIONS:
Locations (36):
- China (36):
  - Anhui Chest Hospital, Hefei, Anhui
  - Peking Union Medical College Hospital, Beijing, Beijing Municipality
  - Chongqing University Cancer Hospital, Chongqing, Chongqing Municipality
  - The First Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality
  - Fujian Cancer Hospital, Fuzhou, Fujian
  - Sun Yat-sen University Cancer Center, Guangzhou, Guangdong
  - The First Affiliated Hospital Sun Yat-Sen University, Guangzhou, Guangdong
  - Yuebei People's Hospital, Shaoguan, Guangdong
  - Affiliated Hospital of Guangdong Medical University, Zhangjiang, Guangdong
  - The Fifth Affiliated Hospital Sun Yat-Sen University, Zhuhai, Guangdong
  - Guangxi Medical University Affiliated Tumor Hospital, Nanning, Guangxi
  - The Fourth Hospital of Hebei medical University, Shijiazhuang, Hebei
  - Henan Cancer Hospital, Zhengzhou, Henan
  - Anyang Cancer Hospital, Anyang, Henang
  - Hubei Cancer Hospital, Wuhan, Hubei
  - Hunan Cancer Hospital, Changsha, Hunan
  - Xiangya Hospital Central South University, Changsha, Hunan
  - The Third Xiangya Hospital of Central South University, Changsha, Hunan
  - Huaian First People's Hospital, Huai'an, Jiangsu
  - Jiangsu Cancer Hospital, Nanjing, Jiangsu
  - Jiangsu People's Hospital, Nanjing, Jiangsu
  - The First Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - Qilu Hospital of Shandong University, Jinan, Shandong
  - Baoji Central Hospital, Baoji, Shanxi
  - Shanxi Cancer Hospital, Taiyuan, Shanxi
  - Xijing Hospital of Airforce Medical University, Xi’an, Shanxi
  - First Affiliated Hospital of Xi'anjiantong University, Xi’an, Shanxi
  - Tianjin Cancer Hospital, Tianjin, Tianjin Municipality
  - The first Hospital of Zhengjiang Province, Hangzhou, Zhejiang
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang
  - Affiliated Hangzhou First People's Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Zhejiang Hospital, Hangzhou, Zhejiang
  - Zhejiang People's Hospital, Hangzhou, Zhejiang
  - Ningbo Medical Center Lihuili Hospital, Ningbo, Zhejiang
  - Taizhou Hospital of Zhejiang Province, Taizhou, Zhejiang
  - Taizhou Central Hospital, Taizhou, Zhejiang

REFERENCES:
- [Derived] Dong B, Chen L, Pang Q, Jiang O, Ge H, Cheng Y, Zhou R, Meng X, Li J, Zhu X, Wang X, Cao Q, Ji Y, Chen M. TQB2450 with or without anlotinib as maintenance treatment in subjects with locally advanced/unresectable non-small cell lung cancer that have not progressed after prior concurrent/sequential chemoradiotherapy (R-ALPS): study protocol for a randomized, double-blind, placebo-controlled, multicenter phase III trial. Transl Lung Cancer Res. 2024 Oct 31;13(10):2828-2837. doi: 10.21037/tlcr-24-362. Epub 2024 Oct 28. PMID 39507039